CLINICAL TRIAL: NCT03086915
Title: Myorelaxation Practice in Paediatric Anesthesia: Retrospective Study
Brief Title: Myorelaxation Practice in Paediatric Anesthesia
Acronym: PAMPE
Status: Completed | Type: Observational
Sponsor: Brno University Hospital (Other)
Collaborators: Masaryk University (Other)
Responsible Party: Principal Investigator, Petr Štourač, MD, doc. MD. Ph.D, Brno University Hospital
Other Study IDs: KDAR FN Brno 3/2017
Record Dates: First submitted 2017-03-05; First posted 2017-03-22 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Neuromuscular Blockade
Keywords: neuromuscular blockade; muscle relaxation; muscle relaxant
MeSH Terms: conditions — Muscle Hypotonia | interventions — Neuromuscular Blocking Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with neuromuscular block: Neuromuscular blocking agent administrated during surgery to the paediatric patient
  Interventions: Drug: Neuromuscular Blocking Agent

INTERVENTIONS:
Drug: Neuromuscular Blocking Agent — Administration of neuromuscular blockers during anesthesia

SUMMARY:
In retrospective data search the investigators will identified the percentage of patients with muscle relaxants administered during perioperative period. The block reversal, typ of drug, percentage of cases with and without reversal will be identified.

DETAILED DESCRIPTION:
The actual percentage of surgeries with the muscle relaxants administered during perioperative period in paediatric patients remain unclear because many surgeries are being performed without muscle relaxation. In this retrospective study, the anesthesiology perioperative data from January 2016 till December 2016 in the tertiary center od Pediatric anesthesia will be searched for the percentage of surgeries with muscle relaxants administered. Type of surgery, age, weight, duration u surgery, muscle relaxants drug and percentage of block reversal will be identified.

ELIGIBILITY:
Inclusion Criteria:

* paediatric patients
* the study period (1/2016-12/2016)
* neuromuscular blocking agent administration during surgery

Exclusion Criteria:

* surgery without neuromuscular blockade

Max Age: 20 Years | Sex: All
Age Groups: Child, Adult
Study Population: Paediatric anesthesiology patients who underwent surgery with neuromuscular blocking agent administered during surgery in tertiary center paediatric anesthesiology department
Sampling Method: Non-Probability Sample
Enrollment: 1650 (Actual)
Dates: Start 2017-03-05 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Percentage of neuromuscular block reversal | 1 year
  The actual percentage of paediatric patients with perioperative neuromuscular blockade with active pharmacology block reversal at the end of surgery

SECONDARY OUTCOMES:
Percentage of surgeries without muscle relaxant administration | 1 year
  Paediatric surgeries without neuromuscular blocking agent administration
Type of neuromuscular blocking agent in paediatric anesthesiology practice | 1 year
  Actual type of neuromuscular blocking agent used in paediatric anesthesiology practice in predefined period.

CONTACTS AND LOCATIONS:
Locations (1):
- Brno University Hospital, Brno, Czechia

IPD SHARING:
Plan to Share IPD: Yes